CLINICAL TRIAL: NCT06286384
Title: Evaluating the Long-term Effects of Microfocused Ultrasound on Facial Tightening Using Quantitative Instruments: Efficacy and Safety
Brief Title: Evaluating the Long-term Effects of Microfocused Ultrasound on Facial Tightening Using Quantitative Instruments
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital of Jinan University (Other)
Responsible Party: Principal Investigator, Hongwei Liu, Plastic Surgery Department Director, First Affiliated Hospital of Jinan University
Other Study IDs: LEMU47
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Facial Aging
Keywords: facial aging; Microfocused Ultrasound; Rejuvenation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A non-randomized, evaluator-blinded study was conducted to observe the changes in the face before and after facial rejuvenation using microfocused ultrasound. The efficacy of microfocused ultrasound in facial rejuvenation was evaluated using standardized photographs in conjunction with a dermatological testing system and to explore the effects of microfocused ultrasound on the function of the skin.

DETAILED DESCRIPTION:
Primary efficacy endpoints:Utilizing the 3D Life Viz mini system for standardized photo modeling enables the comparison and identification of enhancements in treatment outcomes. This research utilized standardized photo modeling to record the facial and mandibular conditions of patients, capturing images both before and after treatment (immediately post-operation and at 7, 30, 90, 180，270 and 360 days). The detection of improvements in treatment effects was then achieved through pairwise comparisons of the modeled data derived from these photographs;Secondary efficacy endpoints: Global Aesthetic Improvement Scale, patient satisfaction scores, Digital Visual Analog Scale

ELIGIBILITY:
Inclusion Criteria:

1. Ages between 25 and 60 years old.
2. Clear manifested skin issues such as sagging and wrinkles: Merz Facial Aesthetics Score of 2 or above.
3. Absence of significant systemic diseases, cardiovascular disorders, impaired liver or kidney function, malignant tumors, etc.
4. Willing to participate in this study and sign an informed consent form.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Individuals with a scar-prone constitution, allergic or abnormally healing skin.
3. Treatment areas with damaged skin, acute inflammation, active infection, rosacea, vitiligo in the progressive stage, or severe acne.
4. Patients with skin conditions such as urticaria, itching, or other dermatological diseases.
5. Those with psychological disorders or drug allergies.
6. Individuals harboring unrealistic expectations about treatment outcomes.
7. Treatment areas containing metal foreign bodies or fillers deemed unsuitable for treatment by the physician.
8. Recent facial laser treatments or injections within the past month, including but not limited to filler treatments such as hyaluronic acid, botulinum toxin, and PRP injection therapy.
9. Any skin-tightening cosmetic treatments on the face or neck within the last three months.
10. Any minimally invasive cosmetic treatments on the face within the last three months.
11. Thread embedding treatments on the face within the last year, excluding thread blepharoplasty.
12. Patients with severe insomnia or those requiring intense sun exposure within the next three months.
13. Patients deemed unsuitable for participation by the investigator.
14. Those unable to cooperate with the treatment and complete all required visits.

Ages: 25 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy women who age naturally
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-07-03 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
Total Volume Change of Nasolabial Folds | before therapy, immediately post-therapy (within 30 minutes), 7 , 30, 90, 180 ,270,and360days
  Utilizing the 3D Life Viz mini system for capturing images both before and after treatment by 30、90、180 days;
Change in Maximum Depth of Nasolabial Folds | before therapy, immediately post-therapy (within 30 minutes), 7 , 30, 90, 180 ,270,and360days
  Utilizing the 3D Life Viz mini system for capturing images both before and after treatment by 30、90、180 days;
Vertical Elevation Value of Nasolabial Fold Curve Projection Curve | before therapy, immediately post-therapy (within 30 minutes), 7 , 30, 90, 180 ,270,and360days
  Utilizing the 3D Life Viz mini system for capturing images both before and after treatment by 30、90、180 days;
Elevation Value of Nasolabial Fold Curve Projection Curve (Along the Nasal Wing Method | before therapy, immediately post-therapy (within 30 minutes), 7 , 30, 90, 180 ,270,and360days
  Utilizing the 3D Life Viz mini system for capturing images both before and after treatment by 30、90、180 days;
Change in Mid-Facial Volume | before therapy, immediately post-therapy (within 30 minutes), 7 , 30, 90, 180 ,270,and360days
  Utilizing the 3D Life Viz mini system for capturing images both before and after treatment by 30、90、180 days;
Brow Lift Height | before therapy, immediately post-therapy (within 30 minutes), 7 , 30, 90, 180 ,270,and360days
  Utilizing the 3D Life Viz mini system for capturing images both before and after treatment by 30、90、180 days;

CONTACTS AND LOCATIONS:
Overall Officials: Hongwei LIU, Study Chair — First Affiliated Hospital of Jinan University
Locations (1):
- First Affiliated Hospital of Jinan University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Li X, Xie G, Yang Z, Li S, Liao X, Lu J, Jiang X, Li K, Xie S, Zhang Z, Xiao L, Huang H, Mao H, Qiao J, Zheng J, Liu H. Evaluating the Long-term Effects of Microfocused Ultrasound on Facial Tightening Using Quantitative Instruments: Efficacy and Safety. Aesthetic Plast Surg. 2025 Sep 10. doi: 10.1007/s00266-025-05205-z. Online ahead of print. PMID 40931143